CLINICAL TRIAL: NCT00283452
Title: Maintaining Physical Activity in Older Adult MCO Members
Brief Title: Keep Active Minnesota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Brian Martinson, PhD, HealthPartners Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 03-024; 1R01AG023410-01 (NIH)
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Physical Activity Maintenance
Keywords: Physical activity maintenance; Interactive phone and mail-based intervention; Older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Participation in phone/mail-based intervention to maintain physical activity.
  Interventions: Behavioral: Phone counseling with written materials
- Control (No Intervention): No intervention; participation in surveys only

INTERVENTIONS:
Behavioral: Phone counseling with written materials — Participation in phone/mail counseling to maintain physical activity
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine whether a new phone and mail based coaching/support program that has been developed is more effective in helping people stay physically active than existing programs that are currently available to all HealthPartners members. We hypothesize that the intervention program will lead to a greater likelihood of physical activity maintenance among moderately active older adults than a usual care condition.

DETAILED DESCRIPTION:
The benefits of physical activity for adults are well established, but less than one-third of older adults in the U.S. have achieved recommended levels of physical activity despite widespread clinical recommendations to increase physical activity in recent years. Clinic-based approaches to increasing physical activity are expensive, difficult to implement in busy practice settings, and have limited reach. Moreover, evidence of the efficacy of such approaches is equivocal. A population based approach may be a more effective and less costly strategy to increase levels of physical activity in older adults. Population studies of physical activity have demonstrated that each year, many sedentary older adults initiate physical activity, but a nearly equal number of those who were active become sedentary. Among older adults initiating physical activity, only half continue to be active 3 months later.

We hypothesize that a population based approach that emphasizes physical activity maintenance can substantially increase physical activity levels in a defined populations of older adults. This hypothesis is tested in a 24-month randomized trial evaluating an innovative, theory-based behavioral intervention to maintain physical activity in a random sample of 50-70 year old adults who have recently become at least moderately active. One thousand (1000) subjects will be randomized to one of two experimental groups: 1) a "usual care" control group, and 2) an interactive phone- and mail-based intervention program tailored to maintaining physical activity in older adults. The primary outcome measures are: 1) physical activity, assessed as kcals/wk expenditure; and 2) physical activity maintenance, assessed as follow-up kcals/wk expenditure relative to baseline. Careful measurement of the penetration of the intervention into a well characterized older adult population, and the costs of the intervention, will be assessed. Psychosocial and behavioral mediators of physical activity maintenance will also be examined.

Study results will be relevant to policy makers, health promotion practitioners and health plans, and will provide practical information on the effectiveness, population penetration, and costs of an intervention designed to maximize population levels of physical activity among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 50 and 70;
* Have HealthPartners insurance for 11 out of the past 12 months;
* Engage in moderate physical activity for a total of 30 minutes at least two days per week;
* Have increased activity level in the past year.

Exclusion Criteria:

* Modified Charlson scores >=3 (calculated using prior year diagnoses);
* Nonskin cancer;
* Congestive heart failure;
* Coronary heart disease;
* Psychotic Illness;
* Substance abuse;
* Terminal illness.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2003-09; Primary Completion 2008-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Absolute level of physical activity: | Assessed at baseline, 6, 12 and 24-month follow-up as kcals/wk expenditure based on survey self-report, validated against activity monitor data in a random sub-sample.
Maintenance of physical activity | Physical activity level relative to baseline assessed at all follow-ups 6, 12, 24 months.

SECONDARY OUTCOMES:
Population penetration: Proportion of those eligible who agree to join the study, and proportion of those randomized to the intervention condition who complete the intervention protocol. | Final endpoint - 24 months
Mediating factors | Level of physical activity self-efficacy, social support for physical activity, and perceived benefits and barriers to activity will also be assessed at baseline and the 6, 12 and 24-month follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C. Martinson, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Senso MM, Anderson CP, Crain AL, Sherwood NE, Martinson BC. Self-reported activity and accelerometry in 2 behavior-maintenance trials. Am J Health Behav. 2014 Mar;38(2):254-64. doi: 10.5993/AJHB.38.2.11. PMID 24629554
- [Derived] Sherwood NE, Martinson BC, Crain AL, Hayes MG, Pronk NP, O'Connor PJ. A new approach to physical activity maintenance: rationale, design, and baseline data from the Keep Active Minnesota Trial. BMC Geriatr. 2008 Jul 25;8:17. doi: 10.1186/1471-2318-8-17. PMID 18655709